CLINICAL TRIAL: NCT00475982
Title: Effect of Weight Loss on Prostate Cancer Pathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CLIN-012-06F
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Prostate Cancer
Keywords: Diet; Insulin-like Growth Factor; Weight Loss
MeSH Terms: conditions — Obesity; Prostatic Neoplasms; Weight Loss

ARMS (2):
- Arm 1: Weight Loss (Experimental): Weight Loss Group
  Interventions: Behavioral: Weight Loss
- Arm 2: No Weight Loss (Active Comparator): No Weight Loss Group
  Interventions: Other: No Weight Loss Group

INTERVENTIONS:
Behavioral: Weight Loss — Subjects undergo a weight loss intervention prior to radical prostatectomy. The intervention includes weekly visits with the dietician, DEXA scanning, blood draws, and anthropometrics.
  Arms: Arm 1: Weight Loss
Other: No Weight Loss Group — These subjects do not undergo a weight loss intervention prior to radical prostatectomy. This group does undergo DEXA scanning, blood draws, and anthropometrics prior to radical prostatectomy.
  Arms: Arm 2: No Weight Loss

SUMMARY:
The purpose of this study is to determine if weight loss prior to radical prostatectomy effects chemical substances in the blood stream and prostate tissue that may affect prostate cancer development and progression.

DETAILED DESCRIPTION:
Obesity is an epidemic, a major public health concern, and is a significant risk factor for progression and mortality from prostate cancer. Prior work in the investigators' laboratory in pre-clinical prostate cancer models and in obese men found that a low fat diet, exercise, and weight loss resulted in antiproliferative and pro-apoptotic effects on prostate cancer tissue through mechanisms related to the IGF-axis. The investigators now propose to conduct a prospective, randomized clinical trial in overweight and obese men with prostate cancer undergoing radical prostatectomy to evaluate if weight loss prior to radical prostatectomy results in antiproliferative and pro-apoptotic effects in prostate cancer tissue. The investigators will accomplish this aim by enrolling overweight and obese men with prostate cancer scheduled to undergo radical prostatectomy. Following informed consent, men will be randomized to either immediate radical prostatectomy or to an 8-week weight loss intervention group that will undergo a diet and exercise weight loss program followed by radical prostatectomy. Proliferation and apoptosis of prostate cancer cells in the prostatectomy specimen will be compared between the groups and relative to the baseline prostate needle biopsy specimens. Further studies will evaluate potential serum surrogate biomarkers that the investigators developed in the investigators' laboratory (ex-vivo serum bioassays) and serum and tissue IGF-axis proteins that have previously been related to obesity, weight loss, and prostate cancer progression. The goal of the investigators' project will be to evaluate the potential anticancer effects of weight loss on prostate cancer tissue and to identify surrogate serum biomarkers that reflect antiproliferative and pro-apoptotic tissue effects and can be applied to future secondary prevention trials in overweight and obese prostate cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Subject is overweight or obese (BMI > 25 kg/m2)
* Patient with pathologically confirmed adenocarcinoma of the prostate and has elected to undergo radical prostatectomy
* Willing to delay radical prostatectomy for 5 to 8-weeks if randomized to the weight loss intervention group.
* Able to adhere to physical activity intervention (able to walk for 30 minutes without rest)
* Able to come to the VA for weight loss visits during the 5 to 8-wk study

Exclusion Criteria:

* Any one of the following: Gleason grade > 4+4, PSA > 20.
* History of ever receiving androgen deprivation therapy, antiandrogen therapy, or finasteride
* Prior prostate radiotherapy (external beam or brachytherapy) or prior cryotherapy
* Diagnosis of diabetes mellitus and on insulin**
* Current use of weight loss medications or enrolled in a diet/weight loss program
* Current use of lycopene supplements*** Significant co-morbidities (i.e. cardiac, pulmonary, liver disease, ongoing alcohol/drug abuse) Cardiac pacemaker

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Aronson, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Weight Loss | Arm 2: No Weight Loss
Started | 23 | 21
Completed | 16 | 18
Not Completed | 7 | 3
Not completed — surgery rescheduled | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Weight Loss | Arm 2: No Weight Loss | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (4.6) | 61.7 (6.6) | 62.5 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 18 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 11 | 15 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 18 | 44

OUTCOME MEASURES:

1. Primary Outcome: Apoptotic Index of the Highest Gleason Grade Malignant Epithelium in the Radical Prostatectomy Specimen Obtained After 8-weeks of the Dietary Intervention
Description: The primary objective is to compare the mean apoptotic index in the radical prostatectomy malignant epithelium between the Weight Loss Group and the Control Group-No Weight Loss. The apoptotic index will be measured in the malignant epithelium with the highest Gleason grade. TUNEL staining was used to identify these apoptotic cells and measure the apoptotic index, which is the percent of cells stained from the sample.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of cells stained
Arm/Group | Arm 1: Weight Loss | Arm 2: No Weight Loss
Number analyzed (Participants) | 16 | 18
percentage of cells stained | 6.9 (10.4) | 5.0 (4.5)
Statistical Analysis 1: Comparison: Arm 1: Weight Loss vs Arm 2: No Weight Loss; Test type: Superiority; p = 0.965, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.965

2. Secondary Outcome: Proliferative Index in Prostate Cancer Epithelium Specimen
Description: The proliferative index in prostate cancer epithelium obtained from the radical prostatectomy specimen. This index was procured by staining the Ki67 protein to measure cell proliferation. (Note: Ki67 is a common indicator of cell proliferation.)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of cells stained
Arm/Group | Arm 1: Weight Loss | Arm 2: No Weight Loss
Number analyzed (Participants) | 16 | 18
percentage of cells stained | 6.69 (5.05) | 5.79 (3)
Statistical Analysis 1: Comparison: Arm 1: Weight Loss vs Arm 2: No Weight Loss; Test type: Superiority; p = 0.884, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.884

3. Secondary Outcome: Change in Serum IGF-related Analytes: IGF-1
Description: This outcome is the measure of the hormone insulin-like growth factor 1 at baseline vs. post-intervention. We measured and compared the concentration (ng/mL) of this hormone.
Time Frame: baseline and post-intervention
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: Weight Loss | Arm 2: No Weight Loss
Number analyzed (Participants) | 16 | 18
ng/mL
  Pre | 165.8 (43.1) | 127.9 (50.7)
  Post | 171.2 (53.4) | 124.8 (53.1)
  Change | 5.38 (19.8) | -3.12 (16.2)
Statistical Analysis 1: Comparison: Arm 1: Weight Loss; intra-analysis within the weight loss arm; Test type: Superiority; p = 0.294, paired t-test
Statistical Analysis 2: Comparison: Arm 2: No Weight Loss; intra-analysis within the control arm; Test type: Superiority; p = 0.440, paired t-test
Statistical Analysis 3: Comparison: Arm 1: Weight Loss vs Arm 2: No Weight Loss; analysis between the weight loss and control arms; Test type: Superiority; p = 0.186, paired t-test; Mean Difference (Net) = 8.49, 95% CI 2-sided [-4.31 to 21.3]

4. Secondary Outcome: Change in Serum IGF-related Analytes: IGFBP-1
Description: This outcome is the measure of the protein, insulin-like growth factor binding protein 1, at baseline vs. post-intervention. We measured and compared the concentration (ng/mL) of this protein.
Time Frame: baseline and post-intervention
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: Weight Loss | Arm 2: No Weight Loss
Number analyzed (Participants) | 16 | 18
ng/mL
  Pre | 8.78 (5.87) | 16.7 (11.1)
  Post | 10.9 (5.77) | 16.6 (11.2)
  Change | 2.19 (5.95) | -0.03 (7.43)
Statistical Analysis 1: Comparison: Arm 1: Weight Loss; intra-analysis within the weight loss arm; Test type: Superiority; p = 0.162, paired t-test
Statistical Analysis 2: Comparison: Arm 2: No Weight Loss; intra-analysis within the control arm; Test type: Superiority; p = 0.986, paired t-test
Statistical Analysis 3: Comparison: Arm 1: Weight Loss vs Arm 2: No Weight Loss; analysis between the weight loss and control arms; Test type: Superiority; p = 0.353, paired t-test; Mean Difference (Net) = 2.22, 95% CI 2-sided [-2.58 to 7.02]

5. Secondary Outcome: Ex-vivo Mitogenic and Apoptotic Activity of Patient Sera on LNCaP Cells
Description: The BRDU assay measures proliferation of cultured cells such as LNCaP. We expose the cells to the patient blood and see if it inhibits prostate cancer cell growth ex vivo. We use optical density (a measure of the amount of light able to pass through the specimen) to indicate the concentration of cell proliferation.
Time Frame: baseline and post-intervention
Measure: Mean (Standard Deviation); unit: density units
Arm/Group | Arm 1: Weight Loss | Arm 2: No Weight Loss
Number analyzed (Participants) | 16 | 18
density units
  Pre | 92.8 (25.8) | 84.8 (27.3)
  Post | 90.8 (23.4) | 83.5 (26.9)
  Change | -2.01 (7.23) | -1.24 (12.72)
Statistical Analysis 1: Comparison: Arm 1: Weight Loss; intra-analysis within the weight loss arm; Test type: Superiority; p = 0.283, paired t-test
Statistical Analysis 2: Comparison: Arm 2: No Weight Loss; intra-analysis within the control arm; Test type: Superiority; p = 0.701, paired t-test
Statistical Analysis 3: Comparison: Arm 1: Weight Loss vs Arm 2: No Weight Loss; analysis between the intervention and control arms; Test type: Superiority; p = 0.835, paired t-test; Mean Difference (Net) = 0.77, 95% CI 2-sided [-6.70 to 8.24]

6. Secondary Outcome: Change in Body Weight
Description: This change in body weight is observed by DEXA, a scanner that measures total body composition.
Time Frame: baseline and post-intervention
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Arm 1: Weight Loss | Arm 2: No Weight Loss
Number analyzed (Participants) | 16 | 18
kg
  Pre | 102.19 (17.15) | 101.02 (17.55)
  Post | 98.47 (16.78) | 99.38 (16.42)
  Change | -3.71 (1.85) | -1.60 (2.32)
Statistical Analysis 1: Comparison: Arm 1: Weight Loss; intra-analysis within the weight loss arm; Test type: Superiority; p = 0.00, paired t-test
Statistical Analysis 2: Comparison: Arm 2: No Weight Loss; intra-analysis within the control arm; Test type: Superiority; p = 0.009, paired t-test
Statistical Analysis 3: Comparison: Arm 1: Weight Loss vs Arm 2: No Weight Loss; analysis between the two arms; Test type: Superiority; p = 0.007, paired t-test; Mean Difference (Net) = 2.11, 95% CI 2-sided [0.64 to 3.59]

7. Secondary Outcome: Change in Percent Body Fat
Description: This change in percent body fat is observed by DEXA, a scanner that measures total body composition.
Time Frame: baseline and post-intervention
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Arm 1: Weight Loss | Arm 2: No Weight Loss
Number analyzed (Participants) | 16 | 18
percentage of body fat
  Pre | 36.8 (3.7) | 36.5 (4.7)
  Post | 35.9 (4.8) | 36.9 (5.4)
  Change | -0.93 (1.92) | 0.41 (0.9)
Statistical Analysis 1: Comparison: Arm 1: Weight Loss; intra-analysis within the weight loss arm; Test type: Superiority; p = 0.073, paired t-test
Statistical Analysis 2: Comparison: Arm 2: No Weight Loss; intra-analysis within the control arm; Test type: Superiority; p = 0.207, paired t-test
Statistical Analysis 3: Comparison: Arm 1: Weight Loss vs Arm 2: No Weight Loss; analysis between the two arms; Test type: Superiority; p = 0.063, paired t-test; Mean Difference (Net) = 1.34, 95% CI 2-sided [-0.08 to 2.75]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Arm 1: Weight Loss | Arm 2: No Weight Loss
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 0/23 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2014-02-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT00475982/Prot_SAP_000.pdf
  • Informed Consent Form: VA GLA ICF (2013-04-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT00475982/ICF_001.pdf
  • Informed Consent Form: UCLA ICF (2011-11-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT00475982/ICF_002.pdf